CLINICAL TRIAL: NCT03349489
Title: Reduction of Basal Insulin to Prevent Hypoglycemia During Exercise in Adults and Adolescents With Type 1 Diabetes Using Insulin Pump Therapy
Brief Title: Insulin-based Strategies to Prevent Hypoglycemia During Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Dr Laurent Legault, MD, FRCP, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RIDE-1 bis
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes; Exercise; Hypoglycemia; Insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Insulin; Insulin Infusion Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduction of insulin basal rate 40 minutes prior to exercise (Active Comparator)
  Interventions: Other: Exercise 2; Device: Dexcom G4 Platinum; Drug: Insulin; Device: Insulin pump
- Reduction of insulin basal rate 90 minutes prior to exercise (Active Comparator)
  Interventions: Other: Exercise 1; Device: Dexcom G4 Platinum; Drug: Insulin; Device: Insulin pump

INTERVENTIONS:
Other: Exercise 1 — Participants will be admitted at the research center at 14:00. At 14:30, participant's insulin basal rate will be reduced by 80%. At 16:00, participants will perform a 60-minute exercise on a stationary bicycle at 60% of their maximal cardiorespiratory capacity (VO2 max). During the exercise period, muscle oxygenation and muscle oxygen extraction will be measure by near infrared spectroscopy. Glucose levels will be measured every 10 minutes during the exercise period. At 17:30, the participant will be discharged.
  Arms: Reduction of insulin basal rate 90 minutes prior to exercise
Other: Exercise 2 — Participants will be admitted at the research center at 14:00. At 15:20, participant's insulin basal rate will be reduced by 80%. At 16:00, participants will perform a 60-minute exercise on a stationary bicycle at 60% of their maximal cardiorespiratory capacity (VO2 max). During the exercise period, muscle oxygenation and muscle oxygen extraction will be measure by near infrared spectroscopy. Glucose levels will be measured every 10 minutes during the exercise period. At 17:30, the participant will be discharged.
  Arms: Reduction of insulin basal rate 40 minutes prior to exercise
Device: Dexcom G4 Platinum — The Dexcom G4 Platinum will be used to measure continuous glucose levels.
Drug: Insulin — Participant's usual fast-acting insulin analog will be used.
Device: Insulin pump — Participant's insulin pump will be used to infuse insulin.

SUMMARY:
It has been reported that insulin basal rate reduction initiated at exercise onset can reduce the hypoglycemic risk during exercise. However, another potentially more efficient strategy to prevent exercise-induced hypoglycemia could be to reduce insulin basal rate a certain time prior to exercise. The objective of this study will be to compare the efficacy of two strategies to prevent exercise-induced hypoglycemia during a 60-minute exercise at moderate intensity: 1) reduce insulin basal rate 40 minutes prior to exercise; 2) reduce insulin basal rate 90 minutes prior to exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 14 years of old.
2. Clinical diagnosis of type 1 diabetes for at least two years.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. Last (less than 2 months) HbA1c ≤ 10%.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Abnormal blood panel and/or anemia.
4. Ongoing pregnancy.
5. Severe hypoglycemic episode within two weeks of screening.
6. Other serious medical illness likely to interfere with study participation or with the ability to complete the exercise periods by the judgment of the investigator (e.g. orthopedic limitation).
7. Failure to comply with team's recommendations (e.g. not willing to change pump parameters, etc.).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in glucose levels | 60 minutes (exercise period)
  Difference between glucose levels at the beginning of the exercise and the lowest glucose levels from the start of the exercise until the end of exercise

SECONDARY OUTCOMES:
Percentage of time of glucose levels spent below 4 mmol/L | 60 minutes (exercise period)
Decremental area under the curve of glucose levels | 60 minutes (exercise period)
Area under the curve of glucose levels < 4 mmol/L | 60 minutes (exercise period)
Number of patients with an exercise-induced hypoglycemia < 3.9 mmol/L | 60 minutes (exercise period)
Number of patients with an exercise-induced hypoglycemia < 3.5 mmol/L | 60 minutes (exercise period)
Number of patients requiring an oral treatment for hypoglycemia | 60 minutes (exercise period)
Total number of hypoglycemia episodes requiring treatment | 60 minutes (exercise period)
Percentage of time of glucose levels spent > 10 mmol/L | 60 minutes (exercise period)
Percentage of time of glucose levels spent between 4-10 mmol/L | 60 minutes (exercise period)
Mean time (minutes) to the first hypoglycemic event | 60 minutes (exercise period)
Amount of carbohydrates needed to treat a hypoglycemic event | 60 minutes (exercise period)
Muscle blood flow | 60 minutes (exercise period)
Percentage of time of glucose levels spent between 4 and 10 mmol/L | 4 hours following end of exercise
Percentage of time of glucose levels spent < 4 mmol/L | 4 hours following end of exercise
Percentage of time of glucose levels spent > 10 mmol/L | 4 hours following end of exercise
Area under the curve of glucose levels < 4 mmol/L | 4 hours following end of exercise
Number of patients requiring an oral treatment for hypoglycemia | 4 hours following end of exercise
Total number of hypoglycemia episodes requiring treatment | 4 hours following end of exercise
Total amount of carbohydrates needed to treat hypoglycemic events | 4 hours following end of exercise
Percentage of time of glucose levels spent between 4 and 10 mmol/L | From the end of exercise period to 6:00 next morning (11 hours)
Percentage of time of glucose levels spent < 4 mmol/L | From the end of exercise period to 6:00 next morning (11 hours)
Percentage of time of glucose levels spent > 10 mmol/L | From the end of exercise period to 6:00 next morning (11 hours)
Area under the curve of glucose levels < 4 mmol/L | From the end of exercise period to 6:00 next morning (11 hours)
Number of patients requiring an oral treatment for hypoglycemia | From the end of exercise period to 6:00 next morning (11 hours)
Total number of hypoglycemia episodes requiring treatment | From the end of exercise period to 6:00 next morning (11 hours)
Total amount of carbohydrates needed to treat hypoglycemic events | From the end of exercise period to 6:00 next morning (11 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Legault, Principal Investigator — Montreal Children's Hospital of the MUHC
Locations (2):
- Canada (2):
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Derived] Tagougui S, Legault L, Heyman E, Messier V, Suppere C, Potter KJ, Pigny P, Berthoin S, Taleb N, Rabasa-Lhoret R. Anticipated Basal Insulin Reduction to Prevent Exercise-Induced Hypoglycemia in Adults and Adolescents Living with Type 1 Diabetes. Diabetes Technol Ther. 2022 May;24(5):307-315. doi: 10.1089/dia.2021.0375. Epub 2022 Apr 27. PMID 35099281